CLINICAL TRIAL: NCT03945513
Title: A Multicenter, Non-Comparative Trial on the Contraceptive Efficacy, Safety, and Tolerability of LPRI-424 (Dienogest 2 mg / Ethinyl Estradiol 0.02 mg) During 13 Cycles
Brief Title: A Multicenter, Non-Comparative Trial on the Contraceptive Efficacy, Safety, and Tolerability of LPRI-424, 13 Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insud Pharma (Industry)
Collaborators: Chemo Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LPRI424/303
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Contraception
Keywords: contraception; hormonal oral contraceptive agents; hormonal oral contraceptive; oral contraceptive
MeSH Terms: interventions — dienogest; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LPRI424 (Experimental): Dienogest 2 mg / ethinyl estradiol 0.02 mg tablet orally once daily for 24 days followed by 4 placebo tablets for a 28 day cycle, for 13 cycles
  Interventions: Drug: LPRI424 (dienogest/ethinylestradiol)

INTERVENTIONS:
Drug: LPRI424 (dienogest/ethinylestradiol) — One LPRI424 tablet once per day for 24 days followed by 4 placebo tablets for 4 days equals one cycle.

SUMMARY:
The main objective of this trial is to demonstrate the contraceptive efficacy of LPRI424, Additional goals of the trial are to demonstrate the safety and tolerability of LPRI424.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, open-label, non-controlled trial in postmenarcheal and premenopausal female subjects, including adolescents, between the ages of 13 and 45 who present to the clinic seeking contraception.

At screening, informed consent will be obtained and the screening procedures will be performed. After confirmation of the subject's eligibility, the subject will be provided with the investigational product and trained in the use of an electronic diary. Afterwards, the subjects will visit the clinical site on Day 20±3 of the 1st, 3rd, 6th and 9th cycles and on Day 29+3 of the 13th cycle. The last clinical site visit will occur 10-14 days after the 13th cycle visit.

The trial will include women who have never used hormonal contraceptives before consent (naïve users), women who have used hormonal contraceptives in the past but have had a contraceptive-free period before consent and a full menstrual cycle during the drug-free period (previous users) as well as women directly switching from another hormonal method (switchers).

Adverse events and safety information will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Sexually active, postmenarcheal and premenopausal female subjects at risk of pregnancy aged between 13-45 years (inclusive) (at the time of trial enrollment).

   Female subjects at risk of pregnancy aged between 13 and 17 years (inclusive) provided that:
   1. Applicable national, state and local laws allow subjects in this age group to consent/assent to receive contraceptive services,
   2. All applicable laws and regulations regarding the informed consent/assent of the subjects to participate in clinical trials are observed.
2. Women who:

   1. have never used hormonal contraceptives before consent/assent (naïve users),
   2. have used hormonal contraceptives in the past, but have had a hormonal contraceptive-free period before consent/assent and a full menstrual cycle during the drug-free period (previous users)
   3. directly switch from another hormonal contraceptive (switchers).
3. Only for subjects who did not use hormonal contraception during the last six months before consent/assent: Regular cycles (i.e. cycle length between 24 and 35 days) during the last six months.
4. At least three complete menstrual cycles after delivery pregnancy (only applicable for women who were pregnant within the last six months).
5. At screening, maximum systolic blood pressure ≤ 140 mm Hg and diastolic blood pressure ≤ 90 mm Hg.
6. Be able and willing to provide written informed consent or assent if the subject is adolescent, prior to undergoing any trial-related procedure.
7. Willing to use trial contraception for thirteen 28-day cycles.
8. Be willing to have intercourse in each cycle of the trial without the need to use back-up contraceptive.
9. Be willing to state that, to her best knowledge, her male sexual partner(s):

   1. Has not had a vasectomy or been previously diagnosed as infertile.
   2. Has not been previously diagnosed or suspected of human immunodeficiency virus (HIV) unless he has subsequently had a negative HIV test.
   3. Has not been known to have engaged in homosexual intercourse in the past five years unless he has had negative HIV test results since then.
   4. Has not shared injection drug needles in the past unless he has had a negative HIV test at least six weeks since last use.
10. Agree not to participate in any other clinical trials during the course of this trial (participation in a non-interventional study is allowed).

Exclusion Criteria:

1. Pregnancy, wish for pregnancy, or breastfeeding subjects.
2. Subject is known to or suspected of not being able to comply with the trial protocol, the use of the trial medication or the use of the trial diary.
3. History of infertility.
4. Abnormal finding on pelvic, breast or ultrasound examination that in the investigator's opinion contraindicates participation in the trial.
5. Unexplained amenorrhea.
6. Known polycystic ovary syndrome (PCOS).
7. Women ≥21 years of age with a Papanicolaou (pap) smear reading low-grade squamous intraepithelial lesion (LGSIL) or higher at screening (or six months prior to screening date). Subjects with atypical squamous cells of undetermined significance (ASC-US) can be included if they are negative for high-risk human papilloma virus (HPV) strains. Subjects <21 years of age do not require a pap smear.
8. Known contraindication or hypersensitivity to ingredients or excipients of the IMP, including:

   1. Presence or risk of a venous thromboembolism (VTE)
   2. Venous thromboembolism - existing VTE (even under treatment with anticoagulants) or history of VTE* (e.g., deep venous thrombosis [DVT] or pulmonary embolism [PE])

      *including a positive family history (VTE ever in a sibling or parent in particular at an age before 50 years)
   3. Known hereditary or acquired predisposition for VTE, e.g., activated protein C (APC) resistance (including Factor V Leiden), antithrombin III deficiency, protein C deficiency, protein S deficiency, or prothrombin-related thrombophilia
   4. Major surgery with prolonged periods of immobilization
   5. High risk of venous thromboembolism due to the presence of multiple risk factors
   6. Presence or risk of an arterial thromboembolism (ATE)
   7. Arterial thromboembolism - existing ATE, history of ATE (e.g., myocardial infarction) or prodromal condition (e.g., angina pectoris)
   8. Cerebrovascular disease - existing stroke, stroke or prodromal disorder (e.g., history of transient ischemic attack [TIA])
   9. Known hereditary or acquired predisposition for ATE, e.g., hyperhomocysteinemia and antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulants)
   10. History of migraine with focal neurological symptoms
   11. High risk of arterial thromboembolism due to multiple risk factors or to the presence of one serious risk factor such as diabetes mellitus with vascular damage, severe hypertension, severe dyslipoproteinemia, smokers or existing or previous pancreatitis, if it is associated with severe hypertriglyceridemia
   12. Existing or previous liver diseases in which liver function has not returned to normal (also Dubin-Johnson and Rotor syndrome)
   13. Existing or previous liver tumors
   14. Known or suspected sex hormone-dependent malignant tumors (e.g., breast or endometrium)
   15. Unexplained vaginal bleeding
   16. Hypersensitivity to the active ingredients or any of the excipients
   17. Concomitant use with the medicinal products containing ombitasvir/paritaprevir/ ritonavir and dasabuvir.
9. Uncontrolled thyroid disorder (i.e., on stable dose of thyroid replacement for less than two months at the time of assent/consent).
10. Uncontrolled concomitant diseases (i.e., not on a stable treatment dose for at least two months at the time of assent/consent).
11. Evidence or history of alcohol, medication or drug abuse (within the last 12 months prior to consent/assent) or medication abuse (within the last three months prior to consent/assent).
12. Predisposition bruising within the last 12 months prior to consent/assent.
13. Known or suspected HIV, hepatitis and/or HPV infection (if the infection is due to aggressive strains) at screening.
14. Less than 3 menses after discontinuing dosing of depot medroxyprogesterone acetate (DMPA or Depo-Provera®) or any combined injectable contraceptive (e.g., Cyclofem®) prior to consent/assent.
15. Long-term treatment (longer than seven consecutive days within a month prior to V1b) of any medication that might interfere with the efficacy of hormonal contraceptives, e.g.:

    1. Anticonvulsants (e.g. phenytoin, carbamazepine, oxcarbazepine, topiramate, felbamate)
    2. Barbiturates (e.g. primidone)
    3. Some antibiotics (such as rifampicin)
    4. HIV medication (such as ritonavir, neviparine and efavirenz)
    5. Bosentan
    6. Griseofulvin
    7. St. John's wort (hypericum perforatum)
    8. Metoclopramide
16. Prohibited medication including the regular intake or use of estrogens, progestogens, activated charcoal, microsomal enzyme-inducing drugs
17. Administration of human chorionic gonadotropin (hCG) or intake of co-medication containing hCG within a month prior to V1b).
18. Progestin-releasing intra-uterine device (IUD) or contraceptive implant received or in place within the last two months prior to consent/assent.
19. Planned regular concomitant use of barrier contraceptive methods, spermicides, IUDs or other contraceptive measures (except occasional use for safety reasons, e.g., to reduce risk of infection).
20. Evidence or history of clinically significant psychiatric illness, such as major depression or schizophrenia, that in the investigator's opinion contraindicates participation in the trialor suicide risk.
21. Planned surgery during the anticipated time of participation in this trial requiring withdrawal of an oral contraceptive.
22. Participation in another trial of an investigational drug or device parallel to the current trial or less than 90 days before consent/assent, or previous participation in the current trial and dispensed trial medication.
23. Subject is a member of the investigator's or sponsor's staff or a relative or family member thereof.
24. Any condition that, in the opinion of the investigator, may jeopardize protocol compliance or the scientific integrity of the trial.
25. Severe COVID-10 disease or less than 3 months after hospitalization due to a COVID-19 disease.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1034 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Number of pregnancies (evaluable cycles) | up to 13 months
  Pearl index (PI) from evaluable cycles in non-breastfeeding women aged ≤ 35 years (at the time of trial enrollment)

SECONDARY OUTCOMES:
Number of pregnancies (all) | up to 13 months
  Pearl Index based on overall cycles (overall PI) in women aged ≤ 35 years (at the time of trial enrollment)
Number of pregnancies (method failures) | up to 13 months
  PI for method failures in women aged ≤ 35 years (at the time of trial enrollment)
Pregnancy ratio | up to 13 months
  Pregnancy ratio in women aged ≤ 35 years (at the time of trial enrollment)
Overall PI, PI for method failures in all women | Up to 13 months
  Overall PI, PI for method failures, PI (using evaluable cycles) and pregnancy ratio (life table analysis) in all women
Overall PI, PI for method failures in women >35 years | Up to 13 months
  5. Overall PI, PI for method failures, PI (using evaluable cycles) and pregnancy ratio (life table analysis) in women aged > 35 years
Number of participants with adverse events as a measure of safety | Up to 13 months
  Adverse events and changes in vital signs, clinical laboratory parameters
Tolerability; Vaginal bleeding pattern | Up to 13 months
  Vaginal bleeding pattern

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Colli, MD, Study Director — Chemo Research
Locations (1):
- Fellows Research Alliance, Inc., Savannah, Georgia, United States